CLINICAL TRIAL: NCT00255489
Title: A Phase I Study of ZD1839 (Iressa) and Palliative Thoracic Radiotherapy in Patients With Non-small Cell Lung Cancer
Brief Title: A Phase I Study of ZD1839 and Palliative Thoracic Radiotherapy in Patients With Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0524
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

INTERVENTIONS:
Drug: Gefitinib
Procedure: palliative thoracic radiotherapy

SUMMARY:
The purpose of this study is to characterize the safety profile of ZD1839 in combination with Palliative thoracic Radiotherapy in patients with non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Patients requiring low dose palliative thoracic irradiation to a field size of less than or equal to 150cm2
* Histologically or cytologically conformed non-small cell lung cancer
* Aged 18 or over

Exclusion Criteria:

* Previous thoracic radiotherapy
* Any condition that may pre-dispose the patient to suffer an individual drug-relaged DLT (dose limiting toxicity) event
* Known hypersensitivity to any component of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2004-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To characterize the safety profile of ZD 1839 in these patients

SECONDARY OUTCOMES:
To measure the quality of life compared to baseline
To measure the change in disease related symptoms compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Iressa Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (2):
- United Kingdom (2):
  - Research Site, Edinburgh
  - Research Site, Leeds